CLINICAL TRIAL: NCT05520749
Title: Efficacy and Safety of Luspatercept in Adult Patients with Transfusion-dependent Anemia Due to Very Low-, Low- and Intermediate-risk (IPSS-R) Myelodysplastic Syndrome with Ring Sideroblasts: a Retrospective Multicenter Study by FISiM-ETS
Brief Title: Efficacy and Safety of Luspatercept: a Study by Fondazione Italiana Sindromi Mielodisplastiche
Acronym: FISiM-Luspa
Status: Completed | Type: Observational
Sponsor: Fondazione Italiana Sindromi Mielodisplastiche-ETS (Other)
Collaborators: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: FISiM-Luspatercept (ICH 3140)
Record Dates: First submitted 2022-08-26; First posted 2022-08-30 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2023-02

CONDITIONS: Myeloid Dysplasia
Keywords: Luspatercept safety; Luspatercept efficacy; Real World Study
MeSH Terms: conditions — Anemia, Refractory, with Excess of Blasts | interventions — luspatercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Luspatercept treated patients: Adult patients (i.e. aged >=18 years) with diagnosis of MDS according to WHO 2016 classification that met IPSS-R criteria for very low, low, or intermediate-risk MDS treated with Luspatercept
  Interventions: Drug: Luspatercept

INTERVENTIONS:
Drug: Luspatercept — Luspatercept treatment in adults with transfusion-dependent anaemia due to MDS

SUMMARY:
Myelodysplastic syndromes (MDS) are a group of malignancies characterized by reduced differentiation and increased apoptosis of hematopoietic progenitor cells, leading to ineffective hematopoiesis. Treatment of MDS varies according to prognosis. Patients with low IPSS-R risk have a low probability of progression to acute myeloid leukemia (AML) and the treatment is aimed at controlling cytopenia and improving quality of life (QOL). Anemia is the most common disease feature, occurring in 80%-85% of low-risk patients, 40% of whom eventually become RBC transfusion-dependent (TD).

Luspatercept is a recombinant fusion protein that selectively binds to ligands belonging to the transforming growth factor-beta (TGF-beta) superfamily. Luspatercept binds to GDF11, GDF8, activin B, and other ligands. This binding leads to inhibition of Smad2/3 signaling, which is abnormally high in disease models of ineffective erythropoiesis such as MDS, resulting in erythroid maturation and differentiation.

Luspatercept is now approved for the treatment of adult patients with TD anemia due to very low-, low-, and intermediate-risk MDS with ring sideroblasts, who had an unsatisfactory response to or are ineligible for erythropoietin-based therapy.

FISiM (Fondazione Italiana Sindromi Mielodidplastiche) promotes a multicenter, retrospective observational study to collect information on the efficacy and safety of luspatercept in a real world Italian population of adult patients with transfusion-dependent anemia due to very low- and intermediate-risk MDS with ring sideroblasts

DETAILED DESCRIPTION:
Myelodysplastic syndromes (MDS) are a group of malignancies characterized by reduced differentiation and increased apoptosis of hematopoietic progenitor cells, leading to ineffective hematopoiesis. The incidence of MDS ranges from 1.5 to 4 cases per 100,000 individuals per year. Prognosis is determined by a number of factors, including age, cytogenetic abnormalities, and cytopenia as determined by the Revised International Prognostic Scoring System (IPSS-R), but also by the occurrence of molecular aberrations (eg, gene mutations) and red blood cell (RBC) transfusion dependence.

Treatment of MDS varies according to prognosis. Patients with low IPSS-R risk have a low probability of progression to acute myeloid leukemia (AML) and the treatment is aimed at controlling cytopenia and improving quality of life (QOL), whereas patients with high-risk disease have a shorter life expectancy and treatment is aimed at modifying the natural course of the disease.

Anemia is the most common disease feature, occurring in 80%-85% of low-risk patients, 40% of whom eventually become RBC transfusion-dependent (TD).

Besides lenalidomide, which is exclusively approved for patients with deletion of chromosome 5q, erythropoiesis-stimulating agents (ESAs) constitute the first option for patients with low risk disease. Patients who do not respond to ESAs have very limited options and ultimately require long-term RBC transfusions. Chronic transfusions lead to secondary iron overload and have a deleterious effect on the patient's QOL.

On April 26, 2019, Celgene Europe BV applied for a marketing authorization via the European Medicines Agency (EMA) centralized procedure for luspatercept (trade name Reblozyl). Luspatercept is a recombinant fusion protein that selectively binds to ligands belonging to the transforming growth factor-beta (TGF-beta) superfamily. Luspatercept binds to GDF11, GDF8, activin B, and other ligands. This binding leads to inhibition of Smad2/3 signaling, which is abnormally high in disease models of ineffective erythropoiesis such as MDS, resulting in erythroid maturation and differentiation.

The review of the benefit-risk balance was conducted by the Committee for Medicinal Products for Human Use (CHMP), and the positive opinion was issued on April 30, 2020. The indication approved in the EU is as follows: "Reblozyl is indicated for the treatment of adult patients with TD anemia due to very low-, low-, and intermediate-risk MDS with ring sideroblasts, who had an unsatisfactory response to or are ineligible for erythropoietin-based therapy.

The clinical development program for luspatercept in MDS consists of 3 clinical trials, including the phase 3, randomized, double-blind, placebo-controlled study ACE-536-MDS-001 (MEDALIST) and 2 supportive phase 2, open-label, single-arm trials (A536-03 and A536-05).

In the MEDALIST trial, adult patients with very low, low, or intermediate IPSS-R risk MDS with ring sideroblasts who required RBC transfusions were randomized 2:1 to luspatercept (1mg/kg) or placebo by the SC route every 3 weeks.16 In both treatment groups, best supportive care could be used when clinically indicated, including RBC transfusions or iron chelation therapy, but excluding ESAs or other MDS-directed agents. The primary endpoint of the trial was the proportion of subjects who were RBC transfusion-independent (RBC-TI) over any 56-day period from week 1 to week 24.

In the MEDALIST trial, 229 subjects very low, low or intermediate IPSS-R risk MDS with ring sideroblasts were randomized: 153 to luspatercept and 76 to placebo (ITT population). Forty-nine (21.4%) patients discontinued from the study, with no differences between arms. Patients' baseline characteristics and prior medication use were well balanced across treatment arms. The percentage of responders (RBC-TI during 56 d through week 24) was 37.91% versus 13.16% (P < 0.0001) for patients receiving luspatercept versus placebo, respectively (Table 1). When the assessment period was extended to 84 days, the proportion of responders was 33.33% versus 11.84% through week 48 and 28.10% versus 7.89% through week 24.

The safety database comprised 571 subjects who received luspatercept. The mean luspatercept treatment duration was 49 weeks (median 45.6). Treatment emergent adverse events (TEAEs) were documented in 95.3% of patients in the pooled luspatercept group, compared to 91.2% of patients in the placebo group. Incidence rates of serious TEAEs (23.8% versus 15.0%), grade ≥3 TEAEs (34.9% versus 25.9%) and TEAEs leading to permanent drug discontinuation (8.8% versus 3.6%) were higher in the pooled luspatercept group. In the MDS cohort, the most frequent TEAEs leading to discontinuation were progression to high-risk MDS, transformation to AML, general physical deterioration and sepsis. Fatal TEAEs were observed in 1.8% versus 2.6% of patients receiving luspatercept versus placebo. The most frequently reported TEAEs (≥15%) in the MDS group were fatigue, diarrhea, nausea, cough, dizziness, hypertension, peripheral edema, headache, viral upper respiratory tract infection, and back pain.

Overall, luspatercept significantly reduced red blood cell (RBC) transfusion requirements in patients with MDS with ring sideroblasts and had a generally manageable tolerability profile in clinical trials. Thus, luspatercept is an emerging treatment option in adults with transfusion-dependent anaemia due to MDS.

Despite that luspatercept is approved based on data of safety and efficacy from a large randomized clinical trial, the authors know that especially for human diseases arising in elderly people, features of subjects included in those randomized trials often do not reflect those of the population in which a therapy is intended to be used. Compliance to treatment and safety in clinical trials can also differ from real world settings. Consequently, in order to drive clinical decision-making process, data from randomized clinical trials should be integrated with evidence generated in a real world setting.

To date, no information is available on the efficacy and safety luspatercept in the treatment of MDS in real world populations. FiSIM (Fondazione Italiana Sindromi Mielodisplastiche) promotes a multicenter, retrospective observational study to collect information on the efficacy and safety of luspatercept in a real world Italian population of adult patients with transfusion-dependent anemia due to very low- and intermediate-risk MDS with ring sideroblasts, who had an unsatisfactory response to or are ineligible for erythropoietin-based therapy.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (i.e. aged >=18 years) with diagnosis of MDS according to WHO 2016 classification that met IPSS-R criteria for very low, low, or intermediate-risk MDS along with the following additional criteria:

* Ring Sideroblasts (RS) ≥15% of erythroid precursors in bone marrow in the absence of SF3B1 mutation, or ≥5% in the presence of SF3B1 mutation;
* Bone marrow blasts <5%;
* Peripheral white blood cell count <13,000/μL;
* ECOG PS 0-2;
* Refractory or intolerant to, or ineligible for prior ESA therapy.
* Required RBC transfusions per the following criteria:
* Mean RBC transfusion requirement ≥2 units/8 weeks in the 16 weeks before the start of luspatercept treatment
* No consecutive 56-day period free from RBCTs in the 16 weeks before the start of luspatercept treatment
* Treatment with luspatercept

Exclusion Criteria:

Any prior treatment with the following therapies:

* Prior therapy with disease modifying agents for MDS including immunomodulatory drugs (eg, lenalidomide), hypomethylating agents (eg, azacitidine or decitabine), and immunosuppressive therapy.
* Presence of the following conditions:
* Pregnancy
* The following blood and laboratory parameters: ANC <500/μL and Platelets <50,000/μL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated with luspatercept in Italy between November 2020 and January 2022 will be included in this study (i.e., around 215 subjects).
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Transfusion independence for 8 weeks or longer during weeks 1 through 24 | From week 1 through week 24 of treatment
  Percentage of patients who achieved RBC Transfusion Independence (RBC-TI) ≥ 8 weeks from week 1 to week 24. RBC-TI response is defined as the absence of any RBC transfusion during any consecutive 56-day (8-week) period (ie, Days 1 to 56, Days 2 to 57, Days 3 to 58, etc.) during the first 24 weeks of study treatment. Patients had to have at least 56 days (≥ 8 weeks) of transfusion independence prior to (and including) the Week 24 date to qualify as a responder. Patients who failed to achieve RBC-TI at least 56 days prior to or on the cut-off date were counted as non-responders.
  Data will be summarised as frequencies and proportions or as medians and range and differences will be estimated by the chi square test (the Fisher exact test when appropriated) or the t test (the Wilcoxon Mann Whitney U test and the ANOVA model when appropriated based on patient characteristics distribution).

SECONDARY OUTCOMES:
Transfusion independence for 12 weeks or longer, assessed during weeks 1 through 24 | From Week 1 through Week 24 of treatment
  Percentage of patients who achieved RBC-TI ≥ 12 weeks from week 1 to week 24. RBC-TI Response is defined as the absence of any RBC transfusion during any consecutive 84-day (12-week) period (ie, Days 1 to 84, Days 2 to 85, Days 3 to 86, etc.) during the first 24 weeks of treatment.
  Data will be summarised as frequencies and proportions or as medians and range and differences will be estimated by the chi square test (the Fisher exact test when appropriated) or the t test (the Wilcoxon Mann Whitney U test and the ANOVA model when appropriated based on patient characteristics distribution).
Transfusion independence for 12 weeks or longer, assessed during weeks 1 through 48 | From Week 1 through Week 48 of treatment
  Percentage of patients who achieved RBC-TI ≥ 12 Weeks from Week 1 to week 48. RBC-TI Response is defined as the absence of any RBC transfusion during any consecutive 84-day (12-week) period (ie, Days 1 to 84, Days 2 to 85, Days 3 to 86, etc.) during the first 48 weeks of treatment.
  Data will be summarised as frequencies and proportions or as medians and range and differences will be estimated by the chi square test (the Fisher exact test when appropriated) or the t test (the Wilcoxon Mann Whitney U test and the ANOVA model when appropriated based on patient characteristics distribution).
Transfusion independence for 8 weeks or longer from week 1 through week 48 | From Week 1 through Week 48 of treatment
  Percentage of patients who achieved RBC-TI ≥ 8 Weeks from week 1 through week 48.
  RBC-TI response is defined as the absence of any RBC transfusion during any consecutive 56-day (8-week) period during the first 48 weeks of study treatment.
  Data will be summarised as frequencies and proportions or as medians and range and differences will be estimated by the chi square test (the Fisher exact test when appropriated) or the t test (the Wilcoxon Mann Whitney U test and the ANOVA model when appropriated based on patient characteristics distribution).

OTHER OUTCOMES:
Erythroid response | Week 1 through 24 or Week 1 Through Week 48
  Percentage of patients who achieved an Hematologic Erythroid Response (HI-E) over any consecutive 56-Day Period.
  A modified HI-E response was defined as the percentage of participants meeting the modified HI-E per the International Working Group (IWG 2018) sustained over 56-day consecutive period during the Treatment period. For patients with a baseline RBC transfusion burden of ≥ 4 units/8 weeks, a HI-E is defined as a reduction in RBC transfusion of at least 4 units/8 weeks; for patients with baseline RBC transfusion burden of <4 units/8 weeks, HI-E is defined as a mean increase in hemoglobin of ≥ 1.5 g/dL for 8 weeks in the absence of RBC transfusions.
Longest duration of primary response (week 1 through week 24) | From start of study treatment to 16 weeks after last dose, up to approximately 93 weeks
  Duration of RBC-TI is defined as the longest duration of response for patients who achieved RBC-TI of ≥ 8 weeks during the treatment period Week 1 through Week 24. Patients who maintained RBC-TI through the end of the treatment period were censored at the date of discontinuation or death, whichever occurred first. Median was estimated from unstratified Kaplan Meier method.
Longest duration of primary response (week 1 through week 48) | From start of study treatment to 16 weeks after last dose, up to approximately 93 weeks
  Duration of RBC-TI is defined as the longest duration of response for patients who achieved RBC-TI of ≥ 8 weeks during the treatment period Week 1 through Week 48. Patients who maintained RBC-TI through the end of the treatment period were censored at the date of discontinuation or death, whichever occurred first. Median was estimated from unstratified Kaplan Meier method.
Mean increase in hemoglobin levels | Week 1 though Week 24 and Week 1 through 48
  Percentage of patients who achieved a Mean Hemoglobin (Hgb) Increase of at Least 1.0 g/dL over any consecutive 56-Day period in absence of RBC Transfusions. A mean hgb increase of ≥ 1.0 g/dL is analyzed as the percentage of patients with a hgb increase ≥1.0 g/dL compared with baseline (after applying the 14/3 day rule) that is sustained over any consecutive 56-day (8-week) period in the absence of RBC transfusions during the treatment period.
Hematologic Improvement in Neutrophil Response | Week 1 through Week 24 or Week 1 Through Week 48 of study treatment
  Percentage of patients who achieved a Hematologic Improvement in Neutrophil Response (HI-N) Over Any Consecutive 56-day Period. Percentage of patients who achieved a hematologic improvement in neutrophil response (HI-N) per IWG criteria sustained over any consecutive 56-day (8-week) period, during the treatment period (Week 1 to Week 24 and Week 1 to Week 48) HI-N was defined as at least a 100% increase and an absolute increase > 0.5 X 10^9/L
Hematologic Improvement in Platelet Response | Week 1 through Week 24 or Week 1 Through Week 48 of study treatment
  Percentage of patients who achieved a Hematologic Improvement in Platelet Response (HI-P) Over Any Consecutive 56-day Period Percentage of patients who achieved a hematologic improvement platelet response (HI-P) was defined as the percentage of participants meeting the HI-P criteria per the IWG sustained over any consecutive 56-day (8-week) period (Week 1 to Week 24 and Week 1 to Week 48) during the treatment period. HI - P response was defined as: Absolute increase of ≥ 30 X 10^9/L in platelets for participants starting with > 20 X 10^9/L platelets; Increase in platelets from < 20 X 10^9/L to > 20 X 10^9/L and by at least 100%
Progression to acute myeloid leukemia | From randomization to study completion (up to approximately 57 months)
  Percentage of patients who progressed to Acute Myeloid Leukemia (AML). Percentage of participants progressing to AML throughout the course of the study
Time to Acute Myeloid Leukemia (AML) Progression | From randomization to study completion (up to approximately 57 months)
  Time to AML progression is defined as the time between randomization date and the first diagnosis of AML as per World Health Organization (WHO) classification of ≥ 20% blasts in peripheral blood or bone marrow. Participants with a diagnosis of AML were considered to have had an event, participants who did not progress to AML at the time of analysis were censored at the last assessment date which did not indicate progression to AML.
Overall Survival | From randomization to study completion (up to approximately 57 months)
  Overall Survival is defined as the time from the date of study drug randomization to death due to any cause. Overall survival was censored at the last date that the participant was known to be alive for participants who were alive at the time of analysis and for those who discontinued from the study or were lost to follow-up.
  Survival curves will be estimated by Kaplan Meier Method and differences between groups will be evaluated by the log-rank test. Hazard ratio and their corresponding 95% confidence intervals will be calculated by the Cox Regression Hazard model. All analyses will be performed using SAS version 9.4.
Mean change in the serum ferritin level | Baseline and Week 9 through Week 24 and Week 33 through Week 48
  Change From Baseline in Mean Serum Ferritin. Mean change from baseline in mean serum ferritin was calculated as the difference of postbaseline mean serum ferritin (averaged over the specified timepoints) and baseline mean serum ferritin.
Safety analyses | From date of first dose up to 42 days after the last dose (up to approximately 83 weeks)
  Number of patients with Treatment Emergent Adverse Events (TEAEs). The outcome measure describes the number of participants who experienced different types of Treatment-emergent adverse events (TEAEs). TEAEs were defined as Adverse Events (AEs) that started on or after the day of the first dose and on or before 42 days after the last dose of luspatercept. The investigator will determine the relationship of an AE to study drug based on the timing of the AE relative to drug administration and whether or not other drugs, therapeutic interventions, or underlying conditions could provide a sufficient explanation for the event. The severity of an AE is evaluated by the investigator according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (Version 4.0) where Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life-threatening and Grade 5 = Death
Change from baseline in RBC Units Transfused over fixed 16-week Period | At Baseline (16 weeks prior to first dose of study treatment) and Weeks 9 to 24 or Weeks 33 to 48
  Mean change in total number of RBC units transfused over a fixed 16-week period (Week 9-24 or Week 33-48) from the total number of RBC units transfused in the 16 weeks immediately on or prior to first dose of study treatment.
Time to Red Blood Cell Transfusion Independence Week 1 Through Week 24 | From first dose to Week 24 of treatment
  Time to Red Blood Cell Transfusion Independence (RBC-TI) - Week 1 Through Week 24. Time to RBC-TI is defined as the time between first dose date and the date of onset of RBC-TI first observed for participants who achieved RBC-TI of ≥ 8 weeks during Week 1 through Week 24
Time to Red Blood Cell Transfusion Independence Week 1 Through Week 48 | From first dose to Week 48 of treatment
  Time to Red Blood Cell Transfusion Independence (RBC-TI) - Week 1 Through Week 48.
  Time to RBC-TI is defined as the time between first dose date and the date of onset of RBC-TI first observed for participants who achieved RBC-TI of ≥ 8 weeks during Week 1 through Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Della Porta, MD, Study Director — Istituto Clinico Humanitas; Valeria Santini, MD, Study Chair — Università degli studi di Firenze - AOU Careggi; Lorenza Borin, MD, Principal Investigator — ASST-MONZA; Daniela Cilloni, MD, Principal Investigator — Aziena Ospedaliera Mauriziano - Torino; Bruno Fattizzo, MD, Principal Investigator — Ospedale Policlinico di Milano; Pellegrino Musto, MD, Principal Investigator — Policlinico di Bari; Esther Oliva, MD, Principal Investigator — Grande Ospedale Metropolitano Bianchi-Melacrino-Morelli di Reggio Calabria; Marta Riva, MD, Principal Investigator — ASST Grande Ospedale Metropolitano Niguarda; Prassede Salutari, MD, Principal Investigator — Presidio Ospedaliero Pescara; Maria Teresa Voso, MD, Principal Investigator — Università Cattolica del Sacro Cuore - Roma
Locations (1):
- Istituto Clinico Humanitas, Milan, Rozzano, Italy

REFERENCES:
- [Derived] Lanino L, Restuccia F, Perego A, Ubezio M, Fattizzo B, Riva M, Consagra A, Musto P, Cilloni D, Oliva EN, Palmieri R, Poloni A, Califano C, Capodanno I, Itri F, Elena C, Fozza C, Pane F, Pelizzari AM, Breccia M, Di Bassiano F, Crisa E, Ferrero D, Giai V, Barraco D, Vaccarino A, Griguolo D, Minetto P, Quintini M, Paolini S, Sanpaolo G, Sessa M, Bocchia M, Di Renzo N, Diral E, Leuzzi L, Genua A, Guarini A, Molteni A, Nicolino B, Occhini U, Rivoli G, Bono R, Calvisi A, Castelli A, Di Bona E, Di Veroli A, Ferrara F, Fianchi L, Galimberti S, Grimaldi D, Marchetti M, Norata M, Frigeni M, Sancetta R, Selleri C, Tanasi I, Tosi P, Turrini M, Giordano L, Finelli C, Pasini P, Naldi I, Santini V, Della Porta MG; Fondazione Italiana Sindromi Mielodisplastiche (FISiM) Clinical network (https://www.fisimematologia.it/). Real-world efficacy and safety of luspatercept and predictive factors of response in patients with lower risk myelodysplastic syndromes with ring sideroblasts. Am J Hematol. 2023 Aug;98(8):E204-E208. doi: 10.1002/ajh.26960. Epub 2023 May 24. No abstract available. PMID 37222267